CLINICAL TRIAL: NCT01510223
Title: Effect of a 5-day Adaptation and Deadaptation Periods to a High-fat Diet Supplemented With Specific Fatty Acids on Gastrointestinal Transit, Appetite and Substrate Utilisation
Brief Title: The Effect of Macronutrients in the Diet on Digestive and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Amir Shafat, Lecturer, Study director,, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NutrientGastEmpt
Record Dates: First submitted 2012-01-05; First posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Obesity; Diabetes; Cardiovascular Diseases
Keywords: Fats; Macronutrients; appetite; gastric emptying; Gastrointestinal transit
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dietary supplementation macademia oil (Experimental): emia oil
  Interventions: Dietary Supplement: Olive oil and macadamia oil; Dietary Supplement: Deadaptation
- Dietary supplementation olive oil (Experimental): Olive oil
  Interventions: Dietary Supplement: Olive oil; Dietary Supplement: Deadaptation
- Dietary Supplementation fish oil (Experimental): fish oil
  Interventions: Dietary Supplement: Olive oil and fish powder; Dietary Supplement: Deadaptation

INTERVENTIONS:
Dietary Supplement: Olive oil — Each volunteer will complete three test trials. The first (CONTROL) and second test trials (HF) were separated by 28 days. The third trial (LF) takes place on the 6th day following the second trial (5 days apart).
  The CON and LF milkshake supplements are identical (272 kcal; 6 g fat). The basic control (CON) or LF milkshake (that the oil was added to) was: 275 g semi skimmed milk, 25 g chocolate milkshake mix, 15 g dried skimmed milk, 1 g xanthan gum. This was made up to 580 ml with still water.
  High-fat milkshake supplements were consumed daily for five days before a test trial. 90 g olive oil added to the supplement for the purpose of the HF intervention phase.
  Other Names: OO
  Arms: Dietary supplementation olive oil
Dietary Supplement: Olive oil and fish powder — Each volunteer will complete three test trials. The first (CONTROL) and second test trials (HF) were separated by 28 days. The third trial (LF) takes place on the 6th day following the second trial (5 days apart).
  The CON and LF milkshake supplements are identical (272 kcal; 6 g fat). The basic control (CON) or LF milkshake (that the oil was added to) was: 275 g semi skimmed milk, 25 g chocolate milkshake mix, 15 g dried skimmed milk, 1 g xanthan gum. This was made up to 580 ml with still water.
  High-fat milkshake supplements were consumed daily for five days before a test trial. 86.67 g olive oil and 3.3 g of n-3 fish powder (500 mg EPA+DHA)added to the supplement for the purpose of the HF intervention phase.
  Other Names: OF
  Arms: Dietary Supplementation fish oil
Dietary Supplement: Olive oil and macadamia oil — Each volunteer will complete three test trials. The first (CONTROL) and second test trials (HF) were separated by 28 days. The third trial (LF) takes place on the 6th day following the second trial (5 days apart).
  The CON and LF milkshake supplements are identical (272 kcal; 6 g fat). The basic control (CON) or LF milkshake (that the oil was added to) was: 275 g semi skimmed milk, 25 g chocolate milkshake mix, 15 g dried skimmed milk, 1 g xanthan gum. This was made up to 580 ml with still water.
  High-fat milkshake supplements were consumed daily for five days before a test trial. 74.82 g olive oil and 15.18 g macadamia nut oil added to the supplement for the purpose of the HF intervention phase.
  Other Names: OM
  Arms: Dietary supplementation macademia oil
Dietary Supplement: Deadaptation — A period of 5 days supplementation with the low-fat milkshake represents a de-adaptation period from high-fat intervention.
  Other Names: DEADAPT

SUMMARY:
This study examined the effect of a 5-day HFD supplemented with specific fatty acids on gastrointestinal transit, appetite, food intake and substrate utilization. Another novel aspect of this chapter was examining whether a subsequent 5-day period was sufficient to reverse the effects of high-fat feeding on the aforementioned parameters.

DETAILED DESCRIPTION:
High-fat (HF) diets of as little as three days have been shown to accelerate GI transit. This study aimed to assess if 5-day HF supplemented diet varying in fatty acid composition were sufficient to accelerate GI transit, appetite responses and substrate utilisation and whether a 5-day deadaptation period to a HF diet would reverse the responses induced by adaptation to a HFD.

The study will be conducted in a randomized, single-blinded manner in 24 healthy subjects. Three 5-day interventions will each followed by a test trial. In the first intervention period (CON), normal diet was supplemented with low-fat (LF) milkshakes (272 kcal, 6 g fat). The second and third interventions will involve repeating previous diet along with HF (1082 kcal, 96 g fat) or LF milkshakes respectively. The three high-fat supplement groups that subjects will be randomized to are as follows: (1) olive oil (90 g oil), (2) olive oil + n-3 EPA/DHA fish powder blend or (3) olive oil + macadamia oil blend.

The effect of 5-day HF diet (daily milkshake supplement: 1082 kcal, 96 g fat) on gastric emptying and mouth to caecum transit time of a high-fat test will be measured using the 13C octanoic acid breath test and H2 inulin breath test respectively for six hours postprandially. During this time course, measurements of subjective appetite sensations by visual analogue scale and substrate utilization by indirect calorimetry were also collected. Subsequently, food intake will be measured using an ad libitum buffet meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-35 years

Exclusion Criteria:

* History of gastrointestinal-related conditions or gastrointestinal disturbance within 3 months of study entry
* diabetes mellitus
* cardiovascular disease
* Allergies to foods in study
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Gastric emptying by 13C octanoic acid breath test | within the first 6.5 hours after ingesting high-fat test meal
  13CO2 breath samples were taken every 15 minutes for six hours. Breath samples for measurement of 13CO2 were analyzed using isotope ratio mass spectrometry and results were expressed relative to Vienna-PeeDee Belemnite. 13CO2 values were expressed as the excess amount in the breath above baseline and converted into moles. This was then fitted to a GE model developed by Ghoos et al. 1993. For all the data, r2 coefficient between the modeled and raw data was calculated and r2 > 0.95. Latency phase (Tlat) and ascension time (Tasc) from Schommartz et al. 1998.

SECONDARY OUTCOMES:
Appetite | Within the first 6.5 hours after a meal
  Satiety was measured using a 150mm VAS to detect changes in hunger, thirst, desire to eat, tiredness, fullness and cold. Variables thirst, tiredness and cold were used to distract volunteers from analysis of their satiety status. This was taken before breakfast, after breakfast, every 30 minutes throughout the six hours and following the buffet meal.
substrate utilization | Within the first 6.5 hours after a meal
  The Douglas Bag technique was employed to collect expired air samples. VO2 and VCO2 were used to calculate substarte oxidation by satndard indirect calorimetry methods.
Food intake by buffet meal | Within 6.5 hours after a meal
  After six hours volunteers were given access to a buffet meal and instructed to eat ad libitum. The buffet meal consisted of a 21 different types of foods and contained a wide variety of foods of varying macronutrient. Foods were covertly weighed before and after presentation and the difference converted to macronutrient intake using food tables or manufacturers' data.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shafat, PhD, Study Director — University of Limerick; Oonagh Markey, BSc, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Limerick, Ireland

REFERENCES:
- [Background] Schommartz B, Ziegler D, Schadewaldt P. Significance of diagnostic parameters in [13C]octanoic acid gastric emptying breath tests. Isotopes Environ Health Stud. 1998;34(1-2):135-43. PMID 9854848
- [Background] Ghoos YF, Maes BD, Geypens BJ, Mys G, Hiele MI, Rutgeerts PJ, Vantrappen G. Measurement of gastric emptying rate of solids by means of a carbon-labeled octanoic acid breath test. Gastroenterology. 1993 Jun;104(6):1640-7. doi: 10.1016/0016-5085(93)90640-x. PMID 8500721